CLINICAL TRIAL: NCT01061151
Title: Breastfeeding Version of the PROMISE Study (Promoting Maternal and Infant Survival Everywhere)
Brief Title: Evaluating Strategies to Reduce Mother-to-Child Transmission of HIV Infection in Resource-Limited Countries
Acronym: PROMISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1077BF (PROMISE); 10777 (Registry Identifier: DAIDS ES); IMPAACT 1077BF; NCT01253538 (obsolete NCT alias)
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: HIV Infections
Keywords: Mother to Child Transmission; HIV Infection; HAART; Maternal Health; Breastfeeding; Perinatal transmission
MeSH Terms: conditions — HIV Infections; Breast Feeding | interventions — Zidovudine; Nevirapine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lamivudine, zidovudine drug combination; Lopinavir

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and outcomes assessor did not receive by-arm tabulations while the study was ongoing.
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Antepartum Arm A (Active Comparator): Mothers received ZDV + sdNVP + TRV Tail
  Interventions: Drug: Zidovudine (ZDV); Drug: Nevirapine (NVP): Antepartum Mothers; Drug: Emtricitabine-tenofovir disoproxil fumarate (Truvada [TRV]) tail; Drug: Nevirapine (NVP): Infant short-course
- Antepartum Arm B (Experimental): Mothers received Triple ARV (3TC-ZDV + LPV-RTV)
  Interventions: Drug: Lamivudine-Zidovudine (3TC-ZDV); Drug: Lopinavir-ritonavir (LPV-RTV); Drug: Nevirapine (NVP): Infant short-course
- Antepartum Arm C (Experimental): Mothers received Triple ARV (TRV + LPV-RTV)
  Interventions: Drug: Lopinavir-ritonavir (LPV-RTV); Drug: Emtricitabine-tenofovir disoproxil fumarate (Truvada [TRV]); Drug: Nevirapine (NVP): Infant short-course
- Late Presenters (Other): Registration to facilitate a structure to screen women and infants for randomization in the Postpartum Component.
  Interventions: Other: No Intervention
- Postpartum Arm A (Maternal Prophylaxis) (Experimental): Mothers received prophylaxis [preferred regimen: TRV + LPV-RTV]. Infants received short-course NVP.
  Interventions: Drug: Lopinavir-ritonavir (LPV-RTV); Drug: Emtricitabine-tenofovir disoproxil fumarate (Truvada [TRV]); Drug: Nevirapine (NVP): Infant short-course
- Postpartum Arm B (Infant Prophylaxis) (Experimental): Infants received extended NVP.
  Interventions: Drug: Nevirapine (NVP): Infant extended
- Maternal Health Arm A (Continue triple ARVs) (Experimental): Mothers continued receiving triple ARV regimen [preferred regimen: TRV + LPV-RTV].
  Interventions: Other: Continue triple ARVs
- Maternal Health Arm B (Discontinue triple ARVs) (Active Comparator): Mothers discontinued triple ARV regimen.
  Interventions: Other: Discontinue triple ARVs

INTERVENTIONS:
Drug: Zidovudine (ZDV) — 300 mg twice daily
  Arms: Antepartum Arm A
Drug: Nevirapine (NVP): Antepartum Mothers — 200 mg at onset of labor
  Arms: Antepartum Arm A
Drug: Emtricitabine-tenofovir disoproxil fumarate (Truvada [TRV]) tail — 200 mg/300 mg x 2 tablets at onset of labor or as soon as possible thereafter; 200 mg/300 mg orally each day after delivery for 7 days or the date of the Week 1 visit (up to 14 days), whichever is later.
  Arms: Antepartum Arm A
Drug: Lamivudine-Zidovudine (3TC-ZDV) — 150 mg/300 mg twice daily
  Arms: Antepartum Arm B
Drug: Lopinavir-ritonavir (LPV-RTV) — 400 mg/100 mg twice daily beginning at >= 14 weeks gestation; 600 mg/150 mg twice daily beginning at >= 28 weeks gestation or at next visit (during third trimester) through delivery; 400 mg/100 mg twice daily after delivery up to 14 days postpartum.
  Arms: Antepartum Arm B; Antepartum Arm C; Postpartum Arm A (Maternal Prophylaxis)
Drug: Emtricitabine-tenofovir disoproxil fumarate (Truvada [TRV]) — 200 mg/300 mg
  Arms: Antepartum Arm C; Postpartum Arm A (Maternal Prophylaxis)
Drug: Nevirapine (NVP): Infant short-course — Oral suspension (dosing according to birth weight) once a day through 42 days of age or through the week 6 visit, whichever is later.
  Arms: Antepartum Arm A; Antepartum Arm B; Antepartum Arm C; Postpartum Arm A (Maternal Prophylaxis)
Drug: Nevirapine (NVP): Infant extended — Oral suspension (dosing according to birth weight) once a day from 6 (up to 14) days of age until there was no longer any risk of MTCT or until the end of follow-up (104 weeks), whichever came first.
  Arms: Postpartum Arm B (Infant Prophylaxis)
Other: No Intervention — Women registered before/during labor received the full Antepartum Arm A regimen.
  Women registered after labor, and who received nevirapine outside of the study, received the Emtricitabine-tenofovir disoproxil fumarate (Truvada [TRV]) tail.
  Arms: Late Presenters
Other: Discontinue triple ARVs — ARVs were discontinued. When protocol specified criteria were met, mothers could be prescribed any licensed antiretroviral medication, as long as the treatment met the definition of HAART (three ARV drugs from two or more drug classes).
  Arms: Maternal Health Arm B (Discontinue triple ARVs)
Other: Continue triple ARVs — Mothers could be prescribed any licensed antiretroviral medication, as long as the treatment met the definition of HAART (three ARV drugs from two or more drug classes).
  Arms: Maternal Health Arm A (Continue triple ARVs)

SUMMARY:
The purpose of this study was to examine, in an integrated and comprehensive fashion, three critical questions currently facing HIV-infected pregnant and postpartum women and their infants:

1. What is the optimal intervention for the prevention of antepartum and intrapartum transmission of HIV?
2. What is the optimal intervention for the prevention of postpartum transmission in breastfeeding (BF) infants?
3. What is the optimal intervention for the preservation of maternal health after the risk period for prevention of mother-to-child-transmission ends (either at delivery or cessation of BF)?

The overall PROMISE protocol had three separate interventional components to address each of these three questions and was conducted at locations in Africa and other parts of the world. Due to variations in the standard of care for HIV-infected pregnant and postpartum women and their infants at different sites, not all of these questions were relevant. Therefore, two separate versions of the PROMISE protocol were developed, each containing only the relevant components. The 1077BF protocol was used at sites where the standard method of infant feeding was breastfeeding, whereas the 1077FF protocol was used at sites where the standard method of infant feeding was formula feeding. The analyses were collapsed across the two protocol versions, and therefore the summaries contain the results of the 1077BF and/or the 1077FF protocols.

DETAILED DESCRIPTION:
The incidence of mother-to-child transmission (MTCT) of HIV has decreased in recent years in the United States, Europe, and other resource-advantaged countries. Several factors have contributed to this decrease, including the administration of HAART during pregnancy, caesarean section delivery methods, and the use of formula instead of breastfeeding to feed infants. However, in resource-limited countries, the incidence of pediatric HIV infection remains high. Many pregnant women in these countries do not receive an adequate course of HAART, and the majority breastfeed their children.

This study was divided into three components (Antepartum, Postpartum, and Maternal Health Components). The following is a description of each of the three open label sequential randomization components, each designed to address one of the following three main objectives:

1. Antepartum Component: This PROMISE component compared the safety and efficacy of different HAART regimens for preventing the transmission of HIV during pregnancy, labor, and delivery.

   * Participants were randomly assigned to one of the following three arms:
   * Maternal Regimens:

     * Arm A : 1) Zidovudine (ZDV) from study entry through delivery, 2) single dose nevirapine (sdNVP) and emtricitabine-tenofovir disoproxil (TRV ) intrapartum, and 3) TRV postpartum for up to 14 days post-partum. Arm A is also labeled as ZDV+sdNVP+TRV tail.
     * Arm B: Lamivudine (3TC)-zidovudine (ZDV) + lopinavir (LPV)-ritonavir (RTV) from study entry up to 14 days postpartum. Arm B is also labeled as 3TC-ZDV/LPV-RTV.
     * Arm C: TRV/LPV-RTV from study entry up to 14 days postpartum. Arm C is also labeled as FTC-TDF/LPV-RTV.
   * All infants born to women enrolled in this study were to receive NVP once a day as soon as possible after birth through 42 days of age or until the Week 6 study visit, whichever was later. Women switched or initiated HAART if it was needed for their own health.
   * During pregnancy, participants attended study visits at study entry, 2 and 4 weeks after entry, and then every 4 weeks until labor and delivery. Women and infants were monitored during labor and delivery and attended a study visit 6 to 14 days after delivery. After delivery, eligibility criteria were assessed for subsequent randomizations (either Postpartum or Maternal Health). If they failed the entry criteria for the subsequent randomization, the mothers remained in follow-up for safety assessments and the infants were followed until the 104 week visit; otherwise they were followed under the subsequent component.
   * All three antepartum arms were not available to all women throughout the PROMISE study. When the trial began, there were limited safety data on tenofovir in pregnancy, and randomization to tenofovir-based ART was limited to women coinfected with HIV and HBV, because benefit was felt to outweigh risk in that group. During period 1 (PROMISE protocol version 2.0 - April 2011 through September 2012), women without HBV coinfection were randomized to either Arm A or Arm B; and Hepatitis B (HBV) co-infected women were randomized to either Arm A, Arm B, or Arm C. However, in October 2012, with increased data on tenofovir in pregnancy, the protocol was modified to allow women regardless of HBV status to be assigned to any of the three regimens during period 2 (PROMISE protocol version 3.0 - October 2012 through the end of antepartum enrollment on October 1, 2014). By arm comparisons were restricted to times in which there were contemporaneous randomizations.
   * Late Presenters: In addition the Antepartum Component, participants could enter PROMISE through the Late Presenters Registration (LP). Late presenters were identified in early or active labor or in the immediate postpartum period (up to 5 days postpartum). The Late Presenters Registration facilitated a structure to screen women and infants for randomization in the Postpartum Component. Women and infants not randomized in the Postpartum Component of PROMISE were followed through the Week 6 visit.
   * There were 3543 mothers and 3407 live born infants enrolled in the Antepartum Component. There were 204 mothers and 204 live born infants in the Late Presenters Registration.
2. Postpartum Component: This PROMISE component compared the safety and efficacy of maternal triple ARV prophylaxis versus daily infant NVP prophylaxis for the prevention of mother-to-child transmission (PMTCT) through breastfeeding. The Postpartum Component consisted of mothers and infants from the Antepartum Component and the Late Presenters Registration who passed the Postpartum Component entry criteria.

   * Participants were randomly assigned to one of two arms:

     * Arm A: Women received LPV-RTV plus TRV from the Week 1 postpartum visit through the end of maternal follow-up (2 to 5 years). Infants received NVP once a day through 42 days of age or until the Week 6 study visit, whichever was later.
     * Arm B: Infants received NVP once a day from the Week 1 postpartum visit until the end of risk for MTCT or until 18 months postpartum (104 weeks). Women did not receive antiretroviral drugs for MTCT prophylaxis.
   * The maternal study visits were at entry, at postpartum weeks 6, 14, 26, and every 12 weeks thereafter. Infant study visits were at entry, every 4 weeks between postpartum weeks 6-26, every 12 weeks between postpartum week 38-98, and at postpartum week 104. At the end of risk for MTCT or 18 months postpartum, the mothers' eligibility criteria were assessed for a subsequent randomization in the Maternal Health Component. If they did not meet entry criteria for the Maternal Health randomization, they remained in follow-up for safety assessments; otherwise they were followed under the Maternal Health Component. Infants were followed until the 104 week visit.
   * Women switched or initiated HAART if it was needed for their own health. If a woman in Arm B initiated HAART then her infant discontinued NVP after 12 weeks of HAART or after her viral load was suppressed, whichever came first.
   * There were 2431 mothers and 2444 infants randomized as part of the Postpartum Component.
3. Maternal Health Component: This PROMISE component randomized women to continue or discontinue HAART after the end of risk for MTCT, either after delivery or after breastfeeding. Participants included women who were receiving the triple ARV regimen in the Postpartum Component; or receiving the triple ARV regimen in the Antepartum Component and were ineligible for the Postpartum Component.

   * Participants were randomly assigned to one of two study arms:

     * Arm A: Participants continued to receive the triple ARV regimen (preferred regimen was LPV-RTV plus TRV).
     * Arm B: Participants discontinued the triple ARV regimen.
   * Study visits occurred at Weeks 4 and 12 and then every 3 months thereafter. Study visits included a medical history review, questionnaires, physical exam, and blood collection. Women switched or initiated a triple ARV regimen if it was needed for their own health.
   * There were 875 mothers randomized as part of the Maternal Health Component.
   * The analyses for the Maternal Health Component we not solely based on the Maternal Health Randomization. Instead there were four prespecified comparison groups for the Maternal Health Component. The four comparison groups used the three randomizations as appropriate to answer the following questions:

     * Question 1: What is the effect on women of using a maternal triple ARV regimen to prevent MTCT during pregnancy, relative to using ZDV + sdNVP + TRV tail to prevent MTCT during pregnancy?
     * Question 2: What is the effect on women of using a maternal triple ARV regimen to prevent MTCT during breastfeeding, relative to using infant NVP to prevent MTCT during breastfeeding?
     * Question 3: What is the effect on women of extending versus discontinuing the antepartum/intrapartum maternal triple ARV regimen at the time of birth?
     * Question 4: What is the effect on women of extending versus discontinuing the postpartum maternal triple ARV regimen after the cessation of risk for MTCT during breastfeeding?
   * There were 1602 mothers included in the analyses for Question 2.

PROMISE mothers were followed for 2 to 5 years, depending on when they enrolled. Infants were followed up to 104 weeks of age. Infant and maternal follow-up ended in September 2016. PROMISE randomizations were halted in the summer of 2014 due to slow accrual to the Later Presenters Registration and the Formula Feeding protocol. Due to the results of an external study, on July 7th 2015 the PROMISE interventions were halted and ART was offered to all participants. Per recommendation from the Data and Safety and Monitoring Board on November 4th 2014, the primary analyses for the Antepartum Component include follow-up through September 10th, 2014. Per recommendation from the Data and Safety and Monitoring Board on November 12th 2015, the primary analyses for the Postpartum Component include follow-up through July 7th, 2015. The Adverse Events in the Reported Adverse Event section include all study follow-up.

ELIGIBILITY:
Antepartum Component Inclusion Criteria:

* Confirmed HIV-1 infection, defined as documented positive results from two samples collected at different time points prior to study entry. More information on this criterion can be found in the protocol.
* Currently pregnant and greater than or equal to 14 weeks gestation based on clinical or other obstetrical measurements
* CD4 count greater than or equal to 350 cells/mm^3, or greater than or equal to the country-specific threshold for initiation of treatment (if that threshold is greater than 350 cells/mm^3), on a specimen obtained within 30 days prior to study entry
* Results of HBV screening (HBsAg testing) available from specimen obtained within 30 days prior to study entry
* The following laboratory values from a specimen obtained within 30 days prior to study entry:

  1. Hemoglobin greater than or equal to 7.5 g/dL
  2. White blood cell count (WBC) greater than or equal to 1,500 cells/mm^3
  3. Absolute neutrophil count (ANC) greater than or equal to 750 cells/mm^3
  4. Platelets greater than or equal to 50,000 cells/mm^3
  5. Alanine aminotransferase (ALT) less than or equal to 2.5 times the upper limit of normal (ULN)
  6. Estimated creatinine clearance of greater than or equal to 60 mL/min using the Cockroft-Gault equation for women
* Plans to deliver in the study-affiliated clinic or hospital
* Has no plans to move outside of the study site area during the 24 months following delivery
* Age of legal majority for the respective country and willing and able to provide written informed consent

Antepartum Component Exclusion Criteria:

* Participation in PROMISE for a prior pregnancy
* Ingestion of any antiretroviral (ARV) regimen with three or more drugs (regardless of duration) or more than 30 days of a single or dual ARV regimen during current pregnancy, according to self report or available medical records
* Requires triple ARV therapy (HAART) for own health based on local standard guidelines
* World Health Organization (WHO) stage 4 disease
* Prior receipt of HAART for maternal treatment indications (e.g., CD4 less than 350 cells/mm^3 or clinical indications); however, could have received ARVs for the sole purpose of prevention of mother-to-child transmission (PMTCT) in previous pregnancies (prior PMTCT regimens could have included a triple ARV regimen, ZDV, 3TC-ZDV, and/or sdNVP for PMTCT, as well as use of a short dual nucleoside reverse transcriptase inhibitor [NRTI] "tail" to reduce risk of NVP resistance.)
* In labor - at onset or beyond (may be eligible for the Late Presenter registration)
* Clinically significant illness or condition requiring systemic treatment and/or hospitalization within 30 days prior to study entry
* Current or history of tuberculosis (TB) disease (positive PPD without TB disease is not exclusionary)
* Use of prohibited medications within 14 days prior to study entry (refer to the protocol for a list of prohibited medications)
* Fetus detected to have serious congenital malformation (ultrasound not required to rule out this condition)
* Current documented conduction heart defect (specialized assessments to rule out this condition are not required; a heart murmur alone and/or type 1 second-degree atrioventricular block [also known as Mobitz I or Wenckebach] is not considered exclusionary)
* Known to meet the local standard criteria for treatment of HBV (Note: HBV DNA testing or other specialized assessments are not expected to be performed as part of this study. A woman would be excluded only if this information is documented from other sources and she meets the local standard criteria for HBV treatment based on those assessments.)
* Social or other circumstances that would hinder long-term follow-up, in the opinion of the site investigator
* Currently incarcerated

Late Presenter Inclusion Criteria:

* Age of legal majority for the respective country
* HIV-1 infection, defined as documented positive results from tests performed on one sample at any time prior to Late Presenter Registration
* In labor (from onset/early labor or beyond) or within 5 days after delivery (with day of delivery considered day 0)
* Has provided written informed consent
* Has no plans to move outside of the study site area during the 24 months following delivery
* If delivered, infant alive and healthy (In the case of a multiple birth, a mother-infant pair will be included in the Late Presenter registration only if both/all infants and the mother meet the eligibility criteria. If only one infant of a multiple birth is alive, the M-I pair may be registered if the infant and the mother otherwise meet all of the eligibility criteria.)

Late Presenter Exclusion Criteria:

* Participation in PROMISE in prior pregnancy
* Ingestion of any antiretroviral regimen during current pregnancy (including for solely for PMTCT), according to self report and available medical records (Note: Use of ARVs provided as standard of care for PMTCT during labor/delivery or postpartum prior to Late Presenter registration is not exclusionary.)
* If known: CD4 count < 350 cells/mm3 or below the country-specific threshold for initiation of treatment, if that threshold is > 350 cells/mm3, on specimen obtained within 30 days prior to study entry (result not required prior to registration)
* Requires triple ARV therapy (HAART) for own health according to local standard guidelines
* WHO Stage 4 disease
* Prior receipt of HAART for maternal treatment indications (e.g., CD4 < 350 cells/mm3 or clinical indications); however, could have received ARVs for the sole purpose of PMTCT in previous pregnancies. (Prior PMTCT regimens could have included a triple ARV regimen, ZDV, 3TCZDV and/or sdNVP for PMTCT, as well as use of a short dual NRTI "tail" to reduce risk of NVP resistance.)
* Current or history of TB disease (positive PPD without TB disease is not exclusionary)
* Known positive infant HIV nucleic acid test (NAT) result (result not required prior to registration)
* Fetal demise or early neonatal death (prior to enrollment/registration)
* Fetus detected with serious congenital malformation (ultrasound not required to rule out this condition)
* Life threatening infant illness or birth condition incompatible with life
* If delivered, infant birth weight < 2.0 kg
* Social or other circumstances which would hinder long-term follow-up, in the opinion of the site investigator
* Current documented conduction heart defect (specialized assessments to rule out this condition are not required; a heart murmur alone and/or type 1 second-degree atrioventricular block (also known as Mobitz I or Wenckebach) is not considered exclusionary)

Postpartum Component Inclusion Criteria:

* Participation in the Antepartum Component or registered as a Late Presenter
* Provided written informed consent
* Has no plans to move outside of the study site area during the 24 months following delivery
* Maternal CD4 count greater than or equal to 350 cells/mm^3, or greater than or equal to the country-specific threshold for initiation of treatment (if that threshold is greater than 350 cells/mm^3), from a specimen obtained within 30 days prior to study entry. More information on this criterion can be found in the protocol.
* The following maternal laboratory values within 30 days prior to entry:

  1. Hemoglobin greater than or equal to 7.0 g/dL
  2. WBC greater than or equal to 1,500 cells/mm^3
  3. ANC greater than or equal to 750 cells/mm^3
  4. Platelets greater than or equal to 50,000 cells/mm^3
  5. ALT less than or equal to 2.5 times the upper limit of normal (ULN)
  6. Estimated creatinine clearance of greater than or equal to 60 mL/min using the Cockroft-Gault equation for women
* Infant alive, healthy, less than or equal to 14 days of age, and uninfected (negative HIV NAT result on specimen drawn prior to study entry)
* The following infant lab values on specimen obtained prior to study entry (within 14 days of birth):

  1. Hemoglobin greater than or equal to 10 g/dL
  2. WBC greater than or equal to 1,500 cells/mm^3
  3. ANC greater than or equal to 750 cells/mm^3
  4. Platelets greater than or equal to 50,000 cells/mm^3
  5. ALT less than or equal to 2.5 times the ULN
* For Registered Late Presenters: Confirmed maternal HIV-1 infection, defined as documented positive results from two samples collected at different time points at any time prior to entry. More information on this criterion can be found in the protocol.

Postpartum Component Exclusion Criteria:

* Positive infant HIV NAT result on specimen drawn prior to entry or no infant HIV NAT result on specimen drawn prior to entry
* Life-threatening infant illness or birth condition incompatible with life
* Infant birth weight less than 2.0 kg
* Social or other circumstances that would hinder long-term follow-up, as judged by the site investigator
* Current or history of TB disease (positive PPD without TB disease is not exclusionary)
* Current documented conduction heart defect (specialized assessments to rule out this condition are not required; a heart murmur alone and/or type 1 second-degree atrioventricular block [also known as Mobitz I or Wenckebach] is not considered exclusionary)
* Requires triple ARV therapy (HAART) for own health

Maternal Health Component Inclusion Criteria:

* Randomly assigned to triple ARV prophylaxis as part of the Postpartum Component and has continued triple ARV prophylaxis until the current randomization without treatment interruption (defined as more than 14 consecutive days of missed dosing) within the previous 30 days; OR randomly assigned to triple ARV prophylaxis in the Antepartum Component but ineligible for the Postpartum Component and has continued triple ARV prophylaxis until the current randomization without treatment interruption (defined as more than 7 consecutive days of missed dosing) within the previous 30 days
* Within two weeks after complete breastfeeding cessation is achieved (defined as completely stopping all exposure to breast milk for greater than or equal to 28 days); i.e., within 29 to 42 days of last breast milk exposure, or reached 18 months postpartum (whichever comes first). Women who reach 18 months postpartum while still breastfeeding will be eligible for entry within 2 weeks before and 4 weeks after the Week 74 visit (Week 72-78); OR if the woman was randomized to triple ARV prophylaxis in the Postpartum Component and her infant is infected and still breastfeeding, she will be eligible for the Maternal Health Component within 42 days of specimen collection for the confirmatory infant HIV NAT; OR if the woman was randomized to triple ARV prophylaxis in the Antepartum Component but mother-infant pair was ineligible for the Postpartum Component she will be eligible for the Maternal Health Component beginning at the Week 1 visit (6-14 days postpartum) through 28 days after delivery; these women should be randomized as soon as possible, ideally within 6-14 days after delivery; OR if the woman was randomized to triple ARV prophylaxis in the Postpartum Component and breastfeeding risk for MTCT ceases for other reasons (e.g., infant death or permanent removal from home through legal services or adoption) within 28 days of event. More information on this criterion can be found in the protocol.
* Provided written informed consent
* CD4 cell count greater than or equal to 350 cells/mm^3, or greater than or equal to the country-specific threshold for initiation of treatment (if that threshold is greater than 350 cells/mm^3), on a specimen obtained within 30 days prior to study entry
* The following laboratory values on a specimen obtained within 30 days prior to study entry:

  1. ANC greater than or equal to 750 cells/mm^3
  2. Hemoglobin greater than or equal to 7.0 gm/dL
  3. Platelet count greater than or equal to 50,000 cells/mm^3
  4. ALT (SGPT) less than or equal to 2.5 times the ULN
  5. Estimated creatinine clearance of greater than or equal to 60 mL/min using the Cockroft-Gault equation for women
* Intend to remain in current geographical area of residence for the duration of study

Maternal Health Component Exclusion Criteria:

* WHO Stage 4 disease
* Clinically significant illness or condition requiring systemic treatment and/or hospitalization within 30 days prior to study entry
* Current or history of TB disease (positive PPD without TB disease is not exclusionary)
* Use of prohibited medications within 14 days prior to study entry
* Social or other circumstances that would hinder long term follow-up as judged by the site investigator
* Current documented conduction heart defect (specialized assessments to rule out this condition are not required; a heart murmur alone and/or type 1 second-degree atrioventricular block [also known as Mobitz I or Wenckebach] is not considered exclusionary)
* Requires a triple ARV regimen for own health

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3747 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Glenn Fowler, MD, MPH, Study Chair — Johns Hopkins Medical Institute, Makerere U.-JHU Research Collaboration
Locations (14):
- Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra, India
- Malawi (2):
  - Blantyre CRS, Blantyre
  - Malawi CRS, Lilongwe
- South Africa (5):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Shandukani Research CRS, Johannesburg, Gauteng
  - Durban Paediatric HIV CRS, Durban, KwaZulu-Natal
  - Umlazi CRS, Durban, KwaZulu-Natal
  - Family Clinical Research Unit (FAM-CRU) CRS, Cape Town, Western Cape
- Kilimanjaro Christian Medical Centre (KCMC), Moshi, Tanzania
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Uganda
- George CRS, Lusaka, Zambia
- Zimbabwe (3):
  - Seke North CRS, Chitungwiza
  - St Mary's CRS, Chitungwiza
  - Harare Family Care CRS, Harare

REFERENCES:
- [Background] Taha T, Nour S, Li Q, Kumwenda N, Kafulafula G, Nkhoma C, Broadhead R. The effect of human immunodeficiency virus and breastfeeding on the nutritional status of African children. Pediatr Infect Dis J. 2010 Jun;29(6):514-8. doi: 10.1097/INF.0b013e3181cda531. PMID 20054287
- [Background] Becquet R, Ekouevi DK, Arrive E, Stringer JS, Meda N, Chaix ML, Treluyer JM, Leroy V, Rouzioux C, Blanche S, Dabis F. Universal antiretroviral therapy for pregnant and breast-feeding HIV-1-infected women: towards the elimination of mother-to-child transmission of HIV-1 in resource-limited settings. Clin Infect Dis. 2009 Dec 15;49(12):1936-45. doi: 10.1086/648446. PMID 19916796
- [Result] U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS. Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0. [Updated August 2009]. Available from: http://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf
- [Result] WHO Case Definitions of HIV for Surveillance and Revised Clinical Staging and Immunological Classification of HIV-related Disease in Adults and Children, World Health Organization, 2007. Available: http://apps.who.int/iris/handle/10665/43699
- [Derived] Bhattacharya D, Tierney C, Butler K, Kiweewa FM, Moodley D, Govender V, Vhembo T, Mohtashemi N, Ship H, Dula D, George K, Chaktoura N, Fowler MG, Peters MG, Currier JS. Comparison of Antiretroviral Therapies in Pregnant Women Living With Human Immunodeficiency Virus and Hepatitis B Virus: A Randomized Controlled Trial. Obstet Gynecol. 2023 Sep 1;142(3):613-624. doi: 10.1097/AOG.0000000000005302. Epub 2023 Aug 3. PMID 37535953
- [Derived] Vhembo T, Baltrusaitis K, Tierney C, Owor M, Dadabhai S, Violari A, Theron G, Moodley D, Mukwasi-Kahari C, George K, Shepherd J, Siberry GK, Browning R, Fowler MG, Stranix-Chibanda L; IMPAACT P1084s study team. Bone and Renal Health in Infants With or Without Breastmilk Exposure to Tenofovir-Based Maternal Antiretroviral Treatment in the PROMISE Randomized Trial. J Acquir Immune Defic Syndr. 2023 Aug 15;93(5):431-437. doi: 10.1097/QAI.0000000000003218. PMID 37199427
- [Derived] Nevrekar N, Butler K, Shapiro DE, Atuhaire P, Taha TE, Makanani B, Chinula L, Owor M, Moodley D, Chipato T, McCarthy K, Flynn PM, Currier J, Fowler MG, Gupta A, Suryavanshi N. Self-reported Antiretroviral Adherence: Association With Maternal Viral Load Suppression in Postpartum Women Living With HIV-1 From Promoting Maternal and Infant Survival Everywhere, a Randomized Controlled Trial in Sub-Saharan Africa and India. J Acquir Immune Defic Syndr. 2023 Jan 1;92(1):76-83. doi: 10.1097/QAI.0000000000003102. Epub 2022 Sep 28. PMID 36170749
- [Derived] Baltrusaitis K, Makanani B, Tierney C, Fowler MG, Moodley D, Theron G, Nyakudya LH, Tomu M, Fairlie L, George K, Heckman B, Knowles K, Browning R, Siberry GK, Taha TE, Stranix-Chibanda L; PROMISE P1084s Study Team. Maternal and infant renal safety following tenofovir disoproxil fumarate exposure during pregnancy in a randomized control trial. BMC Infect Dis. 2022 Jul 20;22(1):634. doi: 10.1186/s12879-022-07608-8. PMID 35858874
- [Derived] Fowler MG, Aizire J, Sikorskii A, Atuhaire P, Ogwang LW, Mutebe A, Katumbi C, Maliwichi L, Familiar I, Taha T, Boivin MJ; PROMISE-NEURODEV study team. Growth deficits in antiretroviral and HIV-exposed uninfected versus unexposed children in Malawi and Uganda persist through 60 months of age. AIDS. 2022 Mar 15;36(4):573-582. doi: 10.1097/QAD.0000000000003122. PMID 34750297
- [Derived] Stranix-Chibanda L, Tierney C, Pinilla M, George K, Aizire J, Chipoka G, Mallewa M, Naidoo M, Nematadzira T, Kusakara B, Violari A, Mbengeranwa T, Njau B, Fairlie L, Theron G, Mubiana-Mbewe M, Khadse S, Browning R, Fowler MG, Siberry GK; PROMISE Study Team. Effect on growth of exposure to maternal antiretroviral therapy in breastmilk versus extended infant nevirapine prophylaxis among HIV-exposed perinatally uninfected infants in the PROMISE randomized trial. PLoS One. 2021 Aug 20;16(8):e0255250. doi: 10.1371/journal.pone.0255250. eCollection 2021. PMID 34415933
- [Derived] Theron G, Brummel S, Fairlie L, Pinilla M, McCarthy K, Owor M, Chinula L, Makanani B, Violari A, Moodley D, Chakhtoura N, Browning R, Hoffman R, Fowler MG. Pregnancy Outcomes of Women Conceiving on Antiretroviral Therapy (ART) Compared to Those Commenced on ART During Pregnancy. Clin Infect Dis. 2021 Jul 15;73(2):e312-e320. doi: 10.1093/cid/ciaa805. PMID 32564058
- [Derived] Aizire J, Sikorskii A, Ogwang LW, Kawalazira R, Mutebe A, Familiar-Lopez I, Mallewa M, Taha T, Boivin MJ, Fowler MG; PROMISE-NEURODEV study team. Decreased growth among antiretroviral drug and HIV-exposed uninfected versus unexposed children in Malawi and Uganda. AIDS. 2020 Feb 1;34(2):215-225. doi: 10.1097/QAD.0000000000002405. PMID 31634154
- [Derived] Hoffman RM, Angelidou KN, Brummel SS, Saidi F, Violari A, Dula D, Mave V, Fairlie L, Theron G, Kamateeka M, Chipato T, Chi BH, Stranix-Chibanda L, Nematadzira T, Moodley D, Bhattacharya D, Gupta A, Coletti A, McIntyre JA, Klingman KL, Chakhtoura N, Shapiro DE, Fowler MG, Currier JS; IMPAACT PROMISE 1077BF/FF team. Maternal health outcomes among HIV-infected breastfeeding women with high CD4 counts: results of a treatment strategy trial. HIV Clin Trials. 2018 Dec;19(6):209-224. doi: 10.1080/15284336.2018.1537327. PMID 30890061
- [Derived] Fowler MG, Qin M, Fiscus SA, Currier JS, Flynn PM, Chipato T, McIntyre J, Gnanashanmugam D, Siberry GK, Coletti AS, Taha TE, Klingman KL, Martinson FE, Owor M, Violari A, Moodley D, Theron GB, Bhosale R, Bobat R, Chi BH, Strehlau R, Mlay P, Loftis AJ, Browning R, Fenton T, Purdue L, Basar M, Shapiro DE, Mofenson LM; IMPAACT 1077BF/1077FF PROMISE Study Team. Benefits and Risks of Antiretroviral Therapy for Perinatal HIV Prevention. N Engl J Med. 2016 Nov 3;375(18):1726-1737. doi: 10.1056/NEJMoa1511691. PMID 27806243
- See also: IMPAACT Study 1077BF — http://www.impaactnetwork.org/studies/1077BF.asp
- See also: MedDra coding of complications — https://www.meddra.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2011 to October 2014, pregnant or just-delivered women were recruited at medical centers in low-income countries.
Groups:
- Antepartum Arm A: Mothers received ZDV+sdNVP+TRV tail
- Antepartum Arm B: Mothers received Triple ARV (3TC-ZDV/LPV-RTV)
- Antepartum Arm C: Mothers received Triple ARV (FTC-TDF/LPV-RTV)
- Late Presenters: Registrational component to assess entry criteria for possible randomization in the Postpartum Component
Period: Protocol Version 2.0: 04/2011-09/2012
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C | Late Presenters
Started | 855 | 861 | 25 | 129
Mothers That Met All Inclusion Criteria | 853 | 861 | 24 | 129
Completed | 623 | 620 | 16 | 101
Not Completed | 232 | 241 | 9 | 28
Not completed — Protocol Violation | 2 | 0 | 0 | 1
Not completed — Death | 6 | 9 | 1 | 2
Not completed — Withdrawal by Subject | 89 | 82 | 2 | 10
Not completed — Lost to Follow-up | 73 | 65 | 2 | 10
Not completed — Site Closure | 15 | 19 | 1 | 0
Not completed — Subject Unable to Get to Clinic | 44 | 61 | 2 | 5
Not completed — Other Reason | 3 | 5 | 1 | 0
Period: Protocol Version 3.0: 10/2012-10/2014
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C | Late Presenters
Started | 694 | 686 | 422 | 75
Mothers That Met All Inclusion Criteria | 694 | 684 | 421 | 75
Completed | 542 | 548 | 345 | 55
Not Completed | 152 | 138 | 77 | 20
Not completed — Protocol Violation | 0 | 0 | 2 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 3 | 5 | 1 | 1
Not completed — Withdrawal by Subject | 54 | 52 | 31 | 3
Not completed — Lost to Follow-up | 49 | 36 | 25 | 4
Not completed — Site Closure | 12 | 11 | 2 | 0
Not completed — Subject Unable to Get to Clinic | 28 | 26 | 15 | 5
Not completed — Other Reason | 5 | 8 | 1 | 3

BASELINE CHARACTERISTICS:
Population: All women in 1077BF/1077FF except those considered ineligible for the analysis after team review.
Groups:
- Total: Total of all reporting groups
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C | Late Presenters | Total
Number analyzed (Participants) | 1547 | 1545 | 445 | 204 | 3741
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26.5 [22.8 to 30.1] | 26.6 [23.3 to 30.3] | 26.4 [22.7 to 30.4] | 26.8 [23.2 to 31.1] | 26.5 [23.0 to 30.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1547 | 1545 | 445 | 204 | 3741
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Non-Hispanic | 1493 | 1487 | 440 | 183 | 3603
  Hispanic (Regardless of Race) | 7 | 12 | 4 | 2 | 25
  Asian, Pacific Islander | 47 | 46 | 1 | 19 | 113
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 489 | 493 | 155 | 31 | 1168
  Tanzania | 23 | 24 | 10 | 0 | 57
  South Africa | 513 | 510 | 78 | 27 | 1128
  Uganda | 207 | 205 | 85 | 9 | 506
  Zimbabwe | 237 | 236 | 99 | 116 | 688
  Zambia | 32 | 31 | 18 | 2 | 83
  India | 46 | 46 | 0 | 19 | 111
Weight [Median (Inter-Quartile Range); unit: kg] — Population: Some late presenters had incomplete measurements
  kg
    number analyzed (Participants) | 1547 | 1545 | 445 | 200 | 3737
    (all) | 64 [57.5 to 73.5] | 64.6 [58 to 74.1] | 64.4 [58 to 75.9] | 60.9 [53 to 68.9] | 64 [57.5 to 74]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Population: Some participants had incomplete measurements for either weight, height, or both.
  kg/m^2
    number analyzed (Participants) | 1545 | 1535 | 442 | 198 | 3720
    (all) | 25.9 [23.5 to 29.5] | 26.3 [23.4 to 29.8] | 26.3 [23.5 to 30.1] | 23.6 [21.8 to 26.8] | 26 [23.4 to 29.6]
HIV RNA level prior to randomization [Median (Inter-Quartile Range); unit: copies/ml] — Population: Baseline HIV RNA data was incomplete for some participants.
  copies/ml
    number analyzed (Participants) | 1540 | 1542 | 445 | 196 | 3723
    (all) | 6409 [1450.5 to 22720] | 8002 [1854 to 28767] | 8393 [1909 to 28454] | 12140 [2407.5 to 39138.5] | 7409 [1708 to 26350]
Viral Load at enrollment [Median (Inter-Quartile Range); unit: log10 copies/mL] — Population: Baseline HIV RNA data was incomplete for some participants.
  log10 copies/mL
    number analyzed (Participants) | 1540 | 1542 | 445 | 196 | 3723
    (all) | 3.8 [3.2 to 4.4] | 3.9 [3.3 to 4.5] | 3.9 [3.3 to 4.5] | 4.1 [3.4 to 4.6] | 3.9 [3.2 to 4.4]
CD4 count at screening [Median (Inter-Quartile Range); unit: cells/mm^3] | 534 [435 to 678] | 526 [439 to 651] | 538 [434 to 684] | 520 [353 to 723] | 530 [434 to 670]
ALT (SGPT) [Median (Inter-Quartile Range); unit: units/liter] — Population: Baseline Alanine Aminotransferase (ALT) values were incomplete for some late presenters.
  units/liter
    number analyzed (Participants) | 1547 | 1545 | 445 | 196 | 3733
    (all) | 12 [10 to 16] | 12 [9 to 15] | 12 [9 to 15] | 16.5 [12 to 22] | 12 [10 to 16]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dl] | 11 [10.2 to 11.8] | 11.1 [10.3 to 11.8] | 11 [10.3 to 11.8] | 10.6 [9.5 to 11.7] | 11 [10.2 to 11.8]
WBC [Median (Inter-Quartile Range); unit: (cells/mm^3)] — Population: Baseline White Blood Cell (WBC) values were incomplete for some participants.
  (cells/mm^3)
    number analyzed (Participants) | 1547 | 1545 | 445 | 196 | 3733
    (all) | 6800 [5670 to 8200] | 6900 [5700 to 8200] | 6840 [5700 to 7900] | 8660 [6895 to 10755] | 6900 [5700 to 8250]
Absolute Neutrophil Count at Baseline [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Baseline Absolute Neutrophil Count (ANC) values were incomplete for some participants.
  cells/mm^3
    number analyzed (Participants) | 1547 | 1545 | 445 | 196 | 3733
    (all) | 4140 [3250 to 5360] | 4209 [3297 to 5300] | 3990 [3220 to 4990] | 5680 [4342.5 to 7662.5] | 4220 [3297 to 5400]
Platelet count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Baseline platelet counts were incomplete for some participants.
  cells/mm^3
    number analyzed (Participants) | 1547 | 1544 | 444 | 195 | 3730
    (all) | 238000 [200000 to 282000] | 236000 [196000 to 282000] | 242500 [203000 to 290000] | 255000 [217000 to 321000] | 239000 [200000 to 285000]
Serum Creatinine [Median (Inter-Quartile Range); unit: mg/dL] — Population: Baseline Serum Creatinine values were incomplete for some participants.
  mg/dL
    number analyzed (Participants) | 1547 | 1545 | 445 | 199 | 3736
    (all) | 0.5 [0.4 to 0.6] | 0.5 [0.4 to 0.6] | 0.5 [0.4 to 0.6] | 0.6 [0.5 to 0.6] | 0.5 [0.4 to 0.6]
WHO Clinical Staging of HIV/AIDS [Count of Participants; unit: Participants] — Clinical staging of HIV/AIDS by WHO definitions (WHO, 2007). Staging is based on clinical findings that guide the diagnosis, evaluation, and management of HIV/AIDS. Clinical stages are categorized as 1 through 4, progressing from primary HIV infection to advanced HIV/AIDS. These stages are defined by specific clinical conditions or symptoms as described in the reference. Population: Baseline WHO staging category was incomplete for some participants.
  Participants
    number analyzed (Participants) | 1544 | 1542 | 445 | 169 | 3700
    Clinical stage I | 1493 | 1506 | 434 | 165 | 3598
    Clinical stage II | 50 | 34 | 11 | 4 | 99
    Clinical stage III | 1 | 2 | 0 | 0 | 3
Calculated Creatinine Clearance (ml/min) [Count of Participants; unit: Participants] — Population: Baseline Calculated Creatinine Clearance values were incomplete for some participants
  Participants
    number analyzed (Participants) | 1547 | 1545 | 445 | 199 | 3736
    <= 50 ml/min | 0 | 0 | 0 | 1 | 1
    > 50 - 60 ml/min | 1 | 0 | 1 | 1 | 3
    > 60 - 80 ml/min | 5 | 5 | 2 | 2 | 14
    > 80 - 100 ml/min | 27 | 31 | 6 | 10 | 74
    > 100 - 120 ml/min | 90 | 108 | 39 | 31 | 268
    > 120 ml/min | 1424 | 1401 | 397 | 154 | 3376
Gestational age at study entry (weeks) [Median (Inter-Quartile Range); unit: weeks] — Population: Baseline gestational age was incomplete for some participants.
  weeks
    number analyzed (Participants) | 1547 | 1544 | 445 | 194 | 3730
    (all) | 25.7 [20.9 to 30.3] | 25.2 [20.6 to 30.1] | 26 [21.9 to 31.1] | 38.6 [37.3 to 40] | 25.6 [21.1 to 30.4]
Gestational age at study entry [Count of Participants; unit: Participants] — Population: Baseline gestational age was incomplete for some participants.
  Participants
    number analyzed (Participants) | 1547 | 1544 | 445 | 10 | 3546
    <14 weeks | 10 | 8 | 2 | 0 | 20
    14 - <28 weeks | 956 | 1008 | 264 | 0 | 2228
    28 - <34 weeks | 418 | 368 | 116 | 1 | 903
    34 - < 37 weeks | 117 | 113 | 45 | 0 | 275
    >= 37 weeks | 46 | 47 | 18 | 9 | 120
The Most Complex ARV Regimen for Prior PMTCT [Count of Participants; unit: Participants] — Population: Baseline ARV history data were incomplete for some participants.
  PI - Protease Inhibitor, NNRTI - Non Nucleoside Reverse Transcriptase Inhibitor, ZDV - Zidovudine, NVP - Nevirapine, NRTI - Nucleoside Reverse Transcriptase Inhibitor
  Participants
    number analyzed (Participants) | 1539 | 1544 | 445 | 204 | 3732
    HAART including NNRTI | 7 | 5 | 2 | 0 | 14
    sdNVP+ZDV | 33 | 48 | 6 | 0 | 87
    sdNVP | 41 | 46 | 15 | 2 | 104
    One PI | 0 | 1 | 0 | 0 | 1
    One NRTI | 2 | 2 | 0 | 0 | 4
    No ARVs for prior PMTCT/no prior pregnancy | 1456 | 1442 | 422 | 202 | 3522
The Last ARV Regimen before Entry during the Current Pregnancy [Count of Participants; unit: Participants] — Population: Baseline ARV history data were incomplete for some participants.
  NNRTI - Non Nucleoside Reverse Transcriptase Inhibitor, NRTI - Nucleoside Reverse Transcriptase Inhibitor, NVP - Nevirapine, ZDV - Zidovudine
  Participants
    number analyzed (Participants) | 1539 | 1544 | 445 | 204 | 3732
    HAART including NNRTI | 1 | 1 | 0 | 7 | 9
    Two NRTIs | 2 | 5 | 3 | 10 | 20
    sdNVP+ZDV | 2 | 0 | 0 | 1 | 3
    sdNVP | 5 | 2 | 0 | 33 | 40
    One NRTI | 326 | 336 | 125 | 0 | 787
    No ARVs during the current pregnancy | 1203 | 1200 | 317 | 153 | 2873

OUTCOME MEASURES:

1. Primary Outcome: Antepartum Component: Number of Confirmed Infant HIV Infections
Description: Defined as HIV nucleic acid test (NAT) positivity of the specimen drawn at either the birth (Day 0-5) or Week 1 (Day 6-14) visit, confirmed by HIV NAT positivity of a second specimen collected at a different time point
Time Frame: Measured at birth or Week 1 study visit
Population: Analysis includes data from periods 1 and 2. Analysis is among the live births with HIV test results summarized for the maternal-infant set (the worst outcome summarized for cases of multiple births). Analysis used the principle of intent to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C
Number analyzed (Participants) | 1386 | 1385 | 325
Participants | 25 | 7 | 2
Statistical Analysis 1: Comparison: Antepartum Arm A vs Antepartum Arm B vs Antepartum Arm C; Arm B and Arm C were combined and compared to Arm A. This comparison was an a priori planned comparison; Test type: Superiority; Risk Difference (RD) = -1.3, 96.5% CI 2-sided [-2.1 to -0.4] — The combination of Arm B and Arm C minus Arm A, based on a repeated confidence interval (Lan-DeMets approach with an O'Brien-Fleming type I error spending function to preserve an experiment-wise type I error rate of 5%)

2. Primary Outcome: Antepartum Component: Number of Mothers With Grade 3 or Higher Toxicities and Selected Grade 2 Hematologic, Renal, and Hepatic Adverse Events
Description: These events were graded using the Division of AIDS (DAIDS) AE Grading Table, Version 1.0, December 2004, Clarification August 2009, which is available on the RSC website (http://rsc.tech-res.com).
Time Frame: Measured through the Week 1 postpartum study visit
Population: Mothers with no safety data available after baseline were not included. Analysis used the principle of intent to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C
Number analyzed (Participants) | 1521 | 1520 | 424
Participants
  Periods 1 and 2: number analyzed (Participants) | 1510 | 1505 | 0
  Periods 1 and 2 | 261 | 318 |
  Period 2: number analyzed (Participants) | 393 | 385 | 380
  Period 2 | 59 | 61 | 60
Statistical Analysis 1: Comparison: Antepartum Arm A vs Antepartum Arm B; Periods 1 and 2; Test type: Superiority; p = 0.008, Fisher Exact
Statistical Analysis 2: Comparison: Antepartum Arm A vs Antepartum Arm C; Period 2; Test type: Superiority; p = 0.77, Fisher Exact
Statistical Analysis 3: Comparison: Antepartum Arm B vs Antepartum Arm C; Period 2; Test type: Superiority; p > 0.99, Fisher Exact

3. Primary Outcome: Antepartum Component: Number of Mothers With Obstetrical Complications
Description: Complications included deaths, diagnoses, signs/symptoms, chemistry lab tests, or hematological lab tests, with grades of 3 (Severe) or worse. Obstetrical complications were those classified by the MedDra coding system as "Pregnancy, puerperium and perinatal conditions", except if the condition was the death of the fetus: "Abortions not specified as induced or spontaneous", "Abortions spontaneous", or "Stillbirth and foetal death."
Time Frame: Measured through the Week 1 postpartum study visit
Population: Mothers who do not have any obstetrical complications information available after study entry are not included. Analysis used the principle of intent to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C
Number analyzed (Participants) | 1521 | 1520 | 424
Participants
  Periods 1 and 2: number analyzed (Participants) | 1521 | 1510 | 0
  Periods 1 and 2 | 89 | 75 |
  Period 2: number analyzed (Participants) | 401 | 398 | 391
  Period 2 | 20 | 12 | 23
Statistical Analysis 1: Comparison: Antepartum Arm A vs Antepartum Arm B; Periods 1 and 2; Test type: Superiority; p = 0.30, Fisher Exact
Statistical Analysis 2: Comparison: Antepartum Arm A vs Antepartum Arm C; Period 2; Test type: Superiority; p = 0.64, Fisher Exact
Statistical Analysis 3: Comparison: Antepartum Arm B vs Antepartum Arm C; Period 2; Test type: Superiority; p = 0.06, Fisher Exact

4. Primary Outcome: Antepartum Component: Number of Mothers With Adverse Pregnancy Outcomes (e.g.,Stillbirth, Preterm Delivery (< 37 Weeks), Low Birth Weight (< 2,500 Grams), and Congenital Anomalies)
Description: Composite outcome
Time Frame: Measured at birth
Population: Includes mothers with confirmed infant birth outcome as live birth, stillbirth, or spontaneous abortion and outcome assessments. Multiple gestation pregnancies (twins and triplets) were summarized at the unique mother level. Analysis used the principle of intent to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C
Number analyzed (Participants) | 1451 | 1447 | 372
Participants
  Periods 1 and 2: number analyzed (Participants) | 1451 | 1447 | 0
  Periods 1 and 2 | 389 | 563 |
  Period 2: number analyzed (Participants) | 349 | 348 | 341
  Period 2 | 91 | 123 | 111
Statistical Analysis 1: Comparison: Antepartum Arm A vs Antepartum Arm B; Periods 1 and 2; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Antepartum Arm A vs Antepartum Arm C; Period 2; Test type: Superiority; p = 0.04, Fisher Exact
Statistical Analysis 3: Comparison: Antepartum Arm B vs Antepartum Arm C; Period 2; Test type: Superiority; p = 0.46, Fisher Exact

5. Primary Outcome: Postpartum Component: Incidence of Confirmed Infant HIV Infection
Description: Defined as infant HIV NAT positivity of a specimen drawn at any post-randomization visit (i.e., any visit after the Week 1 [Day 6-14] visit), confirmed by HIV NAT positivity of a second specimen drawn at a different time point. Analyses were conducted at the Mother-Infant (M-I) pair level, hence the worst outcome for multiple births was counted as a single event.
Time Frame: Measured through site recommended duration of breastfeeding, complete cessation of breastfeeding or 18 months of age, whichever comes first
Population: All Mother-Infant (M-I) pairs, except 1 M-I pair where infant was infected at date of randomization, were included in the analyses. 35 M-I pairs with no post-randomization HIV test results were included and censored at the date of randomization in the analyses. Analyses were intent to treat.
Measure: Number; unit: New cases per 100 person-years
Arm/Group | Postpartum Arm A (Maternal Prophylaxis) | Postpartum Arm B (Infant Prophylaxis)
Number analyzed (Participants) | 1219 | 1211
New cases per 100 person-years | 0.56 | 0.55
Statistical Analysis 1: Comparison: Postpartum Arm A (Maternal Prophylaxis) vs Postpartum Arm B (Infant Prophylaxis); Test type: Superiority; Hazard Ratio (HR) = 1.0, 96% CI 2-sided [0.3 to 3.1] — The confidence interval was based on a repeated confidence interval

6. Primary Outcome: Postpartum Component: Incidence of Grade 3 or Higher Adverse Events and Selected Grade 2 Hematologic, Renal, and Hepatic Adverse Events
Description: as for outcome 2
Time Frame: as for outcome 5
Population: All mothers were included in the analyses. 15 mothers with no post-randomization data were included and censored at the date of randomization in the analyses. Analyses were intent to treat.
Measure: Number; unit: New cases per 100 person-years
Arm/Group | Postpartum Arm A (Maternal Prophylaxis) | Postpartum Arm B (Infant Prophylaxis)
Number analyzed (Participants) | 1220 | 1211
New cases per 100 person-years | 14.4 | 14.1
Statistical Analysis 1: Comparison: Postpartum Arm A (Maternal Prophylaxis) vs Postpartum Arm B (Infant Prophylaxis); Test type: Superiority; p = 0.98, Log Rank

7. Primary Outcome: Maternal Health Component: Incidence of Progression to AIDS-defining Illness or Death
Description: AIDS-defining illness refers to the WHO Clinical Stage 4 illnesses in Appendix IV of the protocol. These events were reviewed and confirmed by an Endpoint review group.
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: This analysis includes mothers on HAART in the Antepartum component and who were eligible and randomized as part of the Postpartum Component or the Maternal Health Component. Analysis used the intent to treat principle.
Measure: Number; unit: New cases per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 797 | 805
New cases per 100 person-years | 0.24 | 0.49
Statistical Analysis 1: Comparison: Maternal Health Arm A (Continue Triple ARVs) vs Maternal Health Arm B (Discontinue Triple ARVs); Test type: Superiority; p = 0.37, Log Rank; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.14 to 2.08] — The hazard ratio compares Arm A relative to Arm B

8. Secondary Outcome: Antepartum Component: Number of Infant HIV Infections
Description: Detected by HIV NAT positivity
Time Frame: Measured at the birth (<= 3 days postpartum) visit
Population: Analysis is among the live births with HIV test results summarized in the maternal-infant set (the worst outcome summarized for multiple births to the same mother). Analysis used the principle of intent to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C
Number analyzed (Participants) | 1386 | 1385 | 325
Participants | 22 | 4 | 2

9. Secondary Outcome: Antepartum Component: Probability of Overall and HIV-free Infant Survival Until 104 Weeks of Age, by Antepartum Arm (in Conjunction With Infants in the Postpartum Component)
Description: For overall survival, failure was defined to be death. For HIV-free survival, failure was defined to be either death or developing HIV. The probability of living, or living without HIV infection, at 104 weeks was calculated by Kaplan-Meier estimation of the survival function.
Time Frame: Measured from birth through 104 weeks of age
Population: Infants in the antepartum component not excluded from analysis; only one infant was included per pregnancy, the one with the earliest failure time. The Periods 1&2 group is infants born to mothers randomized in Arms A and B throughout the PROMISE study (both protocol versions). The period 2 group includes infants born to mothers randomized during the last protocol version only. Since Arm C was only available to all under the last protocol version, this enables unbiased comparison with Arm C.
Measure: Number (95% Confidence Interval); unit: Proportional probability
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C
Number analyzed (Participants) | 1475 | 1459 | 389
Proportional probability
  Overall survival, Periods 1 & 2 group (arms A & B only): number analyzed (Participants) | 1475 | 1459 | 0
  Overall survival, Periods 1 & 2 group (arms A & B only) | 0.959 [0.948 to 0.969] | 0.967 [0.955 to 0.975] |
  Overall survival, period 2 group: number analyzed (Participants) | 404 | 399 | 389
  Overall survival, period 2 group | 0.951 [0.920 to 0.970] | 0.982 [0.962 to 0.991] | 0.942 [0.914 to 0.962]
  HIV-free survival, Periods 1&2 group (arms A&B only): number analyzed (Participants) | 1475 | 1459 | 0
  HIV-free survival, Periods 1&2 group (arms A&B only) | 0.937 [0.923 to 0.948] | 0.947 [0.933 to 0.958] |
  HIV-free survival, period 2 group: number analyzed (Participants) | 404 | 399 | 389
  HIV-free survival, period 2 group | 0.936 [0.903 to 0.958] | 0.940 [0.864 to 0.975] | 0.921 [0.887 to 0.946]
Statistical Analysis 1: Comparison: Antepartum Arm A vs Antepartum Arm B; Overall survival; Test type: Superiority; p = 0.16, Two-sided Z test
Statistical Analysis 2: Comparison: Antepartum Arm A vs Antepartum Arm B; Overall survival, period 2 group; Test type: Superiority; p = 0.0156, Two-sided Z test
Statistical Analysis 3: Comparison: Antepartum Arm A vs Antepartum Arm C; Overall survival, period 2 group; Test type: Superiority; p = 0.31, Two-sided Z test
Statistical Analysis 4: Comparison: Antepartum Arm B vs Antepartum Arm C; Overall survival, period 2 group; Test type: Superiority; p = 0.0022, Two-sided Z test
Statistical Analysis 5: Comparison: Antepartum Arm A vs Antepartum Arm B; HIV-free survival; Test type: Superiority; p = 0.13, Two-sided Z test
Statistical Analysis 6: Comparison: Antepartum Arm A vs Antepartum Arm B; HIV-free survival, period 2 group; Test type: Superiority; p = 0.44, Two-sided Z test
Statistical Analysis 7: Comparison: Antepartum Arm A vs Antepartum Arm C; HIV-free survival, period 2 group; Test type: Superiority; p = 0.24, Two-sided Z test
Statistical Analysis 8: Comparison: Antepartum Arm B vs Antepartum Arm C; HIV-free survival, group 2; Test type: Superiority; p = 0.26, Two-sided Z test

10. Secondary Outcome: Antepartum Component: Maternal HIV RNA Less Than 400 Copies/mL at Delivery
Description: Analysis used the principle of intent to treat.
Time Frame: Measured at the time of delivery
Population: Analysis includes only mothers with HIV RNA data at delivery. Analysis used the principle of intent to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Antepartum Arm A | Antepartum Arm B | Antepartum Arm C
Number analyzed (Participants) | 1547 | 1545 | 445
Participants
  Periods 1 and 2: number analyzed (Participants) | 1344 | 1367 | 0
  Periods 1 and 2: HIV RNA < 400 copies/mL | 415 | 1092 |
  Periods 1 and 2: HIV RNA >= 400 copies/mL | 929 | 275 |
  Period 2: number analyzed (Participants) | 312 | 321 | 304
  Period 2: HIV RNA < 400 copies/mL | 102 | 259 | 225
  Period 2: HIV RNA >= 400 copies/mL | 210 | 62 | 79

11. Secondary Outcome: Postpartum Component: Proportion of Mother-Infant Pairs With no Death or HIV Diagnosis Through 24 Months Post-delivery
Description: Defined as infant HIV NAT positivity of a specimen drawn at any post-randomization visit, confirmed by HIV NAT positivity of a second specimen drawn at a different time point, or infant death. Analyses (Kaplan-Meier probabilities) were conducted at the Mother-Infant (M-I) pair level, hence the worst outcome for multiple births was counted as a single event.
Time Frame: Measured through 24 months post-delivery
Population: All M-I pairs, except 1 M-I pair where infant was infected at date of randomization, were included in the analyses. 3 M-I pairs with no post-randomization data were included and censored at the date of randomization. Analyses were intent to treat.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Postpartum Arm A (Maternal Prophylaxis) | Postpartum Arm B (Infant Prophylaxis)
Number analyzed (Participants) | 1219 | 1211
Probability | 0.971 [0.959 to 0.980] | 0.977 [0.966 to 0.985]

12. Secondary Outcome: Postpartum Component: Proportion of Infants Alive Through 12 and 24 Months Post-delivery
Description: Analyses (Kaplan-Meier probabilities) conducted for all individual infants (rather than M-I pair)
Time Frame: Measured at 12 and 24 months post-delivery
Population: All live-born infants were included in the analyses. 4 infants with no post-randomization data were included and censored at the date of randomization in the analyses. Analyses were intent to treat.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Postpartum Arm A (Maternal Prophylaxis) | Postpartum Arm B (Infant Prophylaxis)
Number analyzed (Participants) | 1227 | 1217
Probability
  12 months post delivery | 0.988 [0.980 to 0.993] | 0.989 [0.981 to 0.994]
  24 months post delivery | 0.978 [0.967 to 0.986] | 0.987 [0.979 to 0.992]

13. Secondary Outcome: Maternal Health Component: Incidence of Death
Description: Number of women who died during the maternal health component; that is, who had been randomized to either continue or discontinue ART after risk of HIV vertical transmission through breastfeeding was over.
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: New cases per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 797 | 805
New cases per 100 person-years | 0.24 [0.18 to 0.32] | 0.43 [0.36 to 0.52]

14. Secondary Outcome: Maternal Health Component: Incidence of AIDS-defining Illness
Description: "AIDS-defining illness" refers to the WHO Clinical Stage 4 illnesses listed in Appendix IV. Stage 4 illnesses were reviewed and confirmed by an Endpoint review group.
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: New cases per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 797 | 805
New cases per 100 person-years | 0.08 [0.05 to 0.12] | 0.25 [0.20 to 0.30]

15. Secondary Outcome: Maternal Health Component: Incidence of HIV/AIDS-related Events
Description: "HIV/AIDS-related event" refers to the WHO Clinical Stage 4 illnesses, pulmonary tuberculosis, and other serious bacterial infections listed in Appendix IV of the protocol. Stage 4 illnesses were reviewed and confirmed by an Endpoint review group.
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: New cases per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 797 | 805
New cases per 100 person-years | 1.14 [0.89 to 1.45] | 1.24 [1.02 to 1.52]

16. Secondary Outcome: Maternal Health Component: Incidence Rate of Cardiovascular or Other Metabolic Events
Description: Cardiovascular or metabolic events of particular concern were included in this analysis. A Poisson model with time to first event as an offset and an over-dispersion parameter was used to estimate incidence rates.
  Metabolic events considered were diabetes mellitus, lipodystrophy, or dyslipidemia. Cardiovascular events considered were hypertension, congestive heart failure, stroke, Transient Ischemia Event (TIA), pulmonary embolism, myocardial infarction (whether acute symptomatic or silent), coronary artery disease, deep vein thrombosis, peripheral vascular disease, or symptomatic HIV-associated cardiomyopathy.
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 794 | 805
events per 100 person-years | 2.9 [2.3 to 3.8] | 5.7 [4.8 to 6.7]

17. Secondary Outcome: Maternal Health Component: Other Targeted Medical Conditions
Description: Other (non-cardiologic) medical conditions of particular concern were included in this outcome. A Poisson model with time to first event as an offset and an over-dispersion parameter was used to estimate incidence rates. Events included were metabolic events, hepatic events, renal events, infections such as pulmonary tuberculosis, malaria, or other serious bacterial infections, and others.
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 794 | 805
events per 100 person-years | 4.0 [3.2 to 4.9] | 4.6 [3.9 to 5.5]

18. Secondary Outcome: Maternal Health Component: Incidence of HIV/AIDS-related Event or Death
Description: as for outcome 15
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: New cases per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 797 | 805
New cases per 100 person-years | 1.30 [1.03 to 1.65] | 1.43 [1.17 to 1.74]

19. Secondary Outcome: Maternal Health Component: Incidence of HIV/AIDS-related Event or World Health Organization (WHO) Clinical Stage 2 or 3 Events
Description: as for outcome 15
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: New cases per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 797 | 805
New cases per 100 person-years | 3.47 [2.80 to 4.31] | 5.61 [4.83 to 6.53]

20. Secondary Outcome: Maternal Health Component: Incidence Rate of Death or Any Condition of Particular Concern
Description: Particular events were targeted as those of particular concern. This outcome considered all such events: death, events defining WHO stages II, III, or IV, targeted cardiovascular adverse events, other targeted adverse events, or cancers which were not AIDS-defining. A complete list can be found in Appendix IV of the Protocol. A Poisson model with time to first event as an offset and an over-dispersion parameter was used to estimate incidence rates.
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 794 | 805
events per 100 person-years | 9.0 [7.3 to 10.9] | 14.0 [12.1 to 16.1]

21. Secondary Outcome: Maternal Health Component: Incidence of Tuberculosis
Description: Incidence of tuberculosis.
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: New cases per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 797 | 805
New cases per 100 person-years | 0.40 [0.32 to 0.51] | 0.31 [0.24 to 0.39]

22. Secondary Outcome: Maternal Health Component: Toxicity: Incidence of Grade 3 or Greater Laboratory Results or Signs and Symptoms and Selected Grade 2 Hematologic, Renal, and Hepatic Laboratory Results
Description: The maternal safety endpoints summarized include grade 2, 3 or 4 hematologies (hemoglobin (Hb), White Blood Cells (WBC), Absolute Neutrophil Count (ANC), platelet count), chemistries (Alanine Aminotransferase (ALT or SGPT), serum creatinine), and grade 3 or 4 signs and symptoms that occurred post-randomization. These events were graded using the Division of AIDS (DAIDS) AE Grading Table, Version 1.0, December 2004, Clarification August 2009, which is available on the RSC website (http://rsc.tech-res.com).
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: New cases per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 797 | 805
New cases per 100 person-years | 15.3 [12.8 to 18.1] | 13.9 [11.9 to 16.3]

23. Secondary Outcome: Maternal Health Component: Incidence Rate of Progression to AIDS-defining Illness, Death, or a Serious Non-AIDS Cardiovascular, Hepatic, or Renal Event
Description: This outcome included AIDS-defining illnesses or cardiovascular, hepatic, or renal adverse events of particular concern which were evaluated as serious. Serious outcomes were both those defined as serious according to the International Conference on Harmonization (ICH) definition, or outcomes with grades equal to or worse than 3 ("Severe"). A Poisson model with time to first event as an offset and an over-dispersion parameter was used to estimate incidence rates. Cardiovascular events considered were hypertension, congestive heart failure, stroke, Transient Ischemia Event (TIA), pulmonary embolism, myocardial infarction (whether acute symptomatic or silent), coronary artery disease, deep vein thrombosis, peripheral vascular disease, or symptomatic HIV-associated cardiomyopathy. Hepatic events considered were cirrhosis and idiopathic sclerosing cholangitis. Renal events considered were renal insufficiency, acute or chronic.
Time Frame: From study entry until July 7, 2015, an average of 94 weeks of follow-up.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Maternal Health Arm A (Continue Triple ARVs) | Maternal Health Arm B (Discontinue Triple ARVs)
Number analyzed (Participants) | 794 | 805
events per 100 person-years | 0.5 [0.4 to 0.6] | 0.9 [0.7 to 1.0]

24. Other Pre Specified Outcome: Maternal Health Component: Cost-effectiveness
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome since cost-effectiveness was not a focus of the study.
Time Frame: From study entry until July 7, 2015.
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Maternal Health Component: Changes in Plasma Concentrations of Inflammatory and Thrombogenic Markers
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome since inflammation and thrombogenic markers were not a focus of the study.
Time Frame: From study entry until July 7, 2015.
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Maternal Health Component: Quality of Life
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome since quality of life was not a focus of the study.
Time Frame: From study entry until July 7, 2015.
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Maternal Health Component: Self-reported Adherence
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome since adherence was not a focus of the study.
Time Frame: From study entry until July 7, 2015.
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Maternal Health Component: Viral Resistance
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome since viral resistance was not a focus of the study.
Time Frame: From study entry until July 7, 2015.
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Postpartum Component: Functional Maternal Antibody and HIV-envelope Binding Responses in Breast Milk and Plasma, Until Cessation of Breastfeeding or 18 Months Postpartum, Whichever Comes First
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome since functional maternal antibody and HIV-envelope binding responses were not a focus of the study.
Time Frame: Measured through the time of cessation of breastfeeding or 18 months postpartum, whichever comes first
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Postpartum Component: Pharmacokinetic Parameters of ARV Drugs Measured in Maternal Plasma, Hair, Breast Milk, and Infant Blood (Plasma or Dried Blood Spot) Samples Collected at Birth; Weeks 1, 6, 14, and 26; and Subsequent Visits During Breastfeeding
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome since pharmacokinetics was not a focus of the study.
Time Frame: Measured through the last study visit during breastfeeding, or 18 months postpartum, whichever comes first
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Postpartum Component: Cost-effectiveness and Feasibility of the Study ARV Prophylaxis Regimens
Description: as for outcome 24
Time Frame: Measured at the end of the 5-year study period
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Postpartum Component: Rates and Patterns of Maternal and Infant Resistance to the Maternal and Infant ARV Regimens
Description: as for outcome 28
Time Frame: Measured at the end of the 5-year study period
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Postpartum Component: Adherence to the Maternal and/or Infant ARV Regimens, as Measured by Maternal Report and Hair Measures
Description: Adherence is by maternal report; adherence through hair analysis is not included here.
  The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome since adherence was not a focus of the study.
Time Frame: Week 6 visit (14 days - 9 weeks postpartum); Week 14 visit (10-19 weeks postpartum); Week 26 visit (20 to 31 weeks postpartum); Week 50 visit (44 to 55 weeks postpartum); and Week 74 visit (68 to 80 weeks postpartum).
Population: Women or infants in the postpartum component who had been included in the primary efficacy analysis (outcome measure #5 above), i.e., who had not yet reached the site recommended duration of breastfeeding, complete cessation of breastfeeding or 18 months of age, whichever comes first, and whose adherence questionnaire was filled out.
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Arm A (Maternal Prophylaxis) | Postpartum Arm B (Infant Prophylaxis)
Number analyzed (Participants) | 1220 | 1211
Participants
  Week 6 visit: number analyzed (Participants) | 1172 | 1182
  Week 6 visit: Never missed a dose | 1003 | 1104
  Week 6 visit: Missed dose over 1 month ago | 12 | 0
  Week 6 visit: Missed dose 2-4 weeks ago | 17 | 4
  Week 6 visit: Missed dose within last 2 weeks | 140 | 74
  Week 14 visit: number analyzed (Participants) | 1123 | 1140
  Week 14 visit: Never missed a dose | 956 | 1081
  Week 14 visit: Missed dose over 1 month ago | 20 | 0
  Week 14 visit: Missed dose 2-4 weeks ago | 35 | 9
  Week 14 visit: Missed dose within last 2 weeks | 112 | 50
  Week 26 visit: number analyzed (Participants) | 1070 | 1091
  Week 26 visit: Never missed a dose | 888 | 1035
  Week 26 visit: Missed dose over 1 month ago | 48 | 1
  Week 26 visit: Missed dose 2-4 weeks ago | 31 | 8
  Week 26 visit: Missed dose within last 2 weeks | 103 | 47
  Week 50 visit: number analyzed (Participants) | 851 | 887
  Week 50 visit: Never missed a dose | 716 | 841
  Week 50 visit: Missed dose over 1 month ago | 37 | 9
  Week 50 visit: Missed dose 2-4 weeks ago | 34 | 7
  Week 50 visit: Missed dose within last 2 weeks | 64 | 30
  Week 74 visit: number analyzed (Participants) | 377 | 389
  Week 74 visit: Never missed a dose | 311 | 377
  Week 74 visit: Missed dose over 1 month ago | 15 | 2
  Week 74 visit: Missed dose 2-4 weeks ago | 17 | 1
  Week 74 visit: Missed dose within last 2 weeks | 34 | 9

34. Other Pre Specified Outcome: Antepartum Component: Antepartum Change in HBV DNA Viral Load Between Week 8 and Baseline Levels (Using Log HBV DNA) Among Women With Detectable HBV DNA Viral Loads at Baseline and Other HBV Outcome Measures
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome measure since changes in HBV DNA Viral Load was not a focus of the study.
Time Frame: Measured at Week 8
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Antepartum Component: Cost Effectiveness and Feasibility of the Trial ARV Regimens
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome measure since cost effectiveness was not a focus of the study.
Time Frame: Measured at the end of the 5-year study period
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Antepartum Component: Maternal and Infant Viral Resistance to the Maternal and Infant ARV Strategies
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome measure since viral resistance was not a focus of the study.
Time Frame: Measured at the end of the 5-year study period
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Antepartum Component: Adherence to the Maternal Antiretroviral (ARV) Regimen, as Measured by Maternal Report
Description: The protocol did not distinguish between outcomes essential to the primary publication and outcomes for subsequent publications of lesser priority. This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome measure since adherence was not a focus of the study.
Time Frame: Measured through the Week 1 postpartum study visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study entry (for mothers) or birth (for infants) until study completion on September 30, 2016, an average of 169 weeks for mothers and through 24 months or September 30, 2016 for infants, whichever came first.
Description: Some women lost their infant before delivery. Expedited adverse event (AE) reporting followed Intensive Division of AIDS (DAIDS) Reporting Level, which included AEs resulting in death, congenital anomalies, fetal losses, significant disabilities requiring hospitalization and all grade 2 and higher hematology or chemistry events and grade 3 or 4 sign or symptoms. These events were graded using the DAIDS AE Grading Table, Version 1.0, 2009, available on the RSC website (http://rsc.tech-res.com).
Groups:
- Mother, (AP) ZDV+sdNVP+TRV Tail; Infant, (Mother Received ZDV+sdNVP+TRV Tail): Mothers received ZDV+sdNVP+TRV tail
- Mother, (AP) Triple ARV (3TC-ZDV/LPV-RTV); Infant, (Mother Received Triple ARV (3TC-ZDV/LPV-RTV)): Mothers received Triple ARV (3TC-ZDV/LPV-RTV)
- Mother, (AP) Triple ARV (FTC-TDF/LPV-RTV); Infant, (Mother Received Triple ARV (FTC-TDF/LPV-RTV)): Mothers received Triple ARV (FTC-TDF/LPV-RTV)
- Mother, LP; Infant, LP: Registrational component to assess entry criteria for possible randomization in the Postpartum Component
Arm/Group | Mother, (AP) ZDV+sdNVP+TRV Tail | Mother, (AP) Triple ARV (3TC-ZDV/LPV-RTV) | Mother, (AP) Triple ARV (FTC-TDF/LPV-RTV) | Mother, LP | Infant, (Mother Received ZDV+sdNVP+TRV Tail) | Infant, (Mother Received Triple ARV (3TC-ZDV/LPV-RTV)) | Infant, (Mother Received Triple ARV (FTC-TDF/LPV-RTV)) | Infant, LP
All-Cause Mortality (participants affected / at risk) | 9/1547 | 14/1545 | 2/445 | 3/204 | 59/1500 | 46/1478 | 27/429 | 5/204
Serious Adverse Events (participants affected / at risk) | 267/1547 | 276/1545 | 69/445 | 10/204 | 296/1500 | 287/1478 | 113/429 | 20/204
Other Adverse Events (participants affected / at risk) | 1413/1547 | 1414/1545 | 388/445 | 169/204 | 1406/1500 | 1388/1478 | 403/429 | 170/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mother, (AP) ZDV+sdNVP+TRV Tail (N=1547) | Mother, (AP) Triple ARV (3TC-ZDV/LPV-RTV) (N=1545) | Mother, (AP) Triple ARV (FTC-TDF/LPV-RTV) (N=445) | Mother, LP (N=204) | Infant, (Mother Received ZDV+sdNVP+TRV Tail) (N=1500) | Infant, (Mother Received Triple ARV (3TC-ZDV/LPV-RTV)) (N=1478) | Infant, (Mother Received Triple ARV (FTC-TDF/LPV-RTV)) (N=429) | Infant, LP (N=204)
Anaemia (Blood and lymphatic system disorders) | 13 | 16 | 4 | 3 | 10 | 11 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 4 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cleft palate (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Congenital anaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Congenital anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Congenital genital malformation male (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Congenital malaria (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Congenital megacolon (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Congenital musculoskeletal anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Congenital pneumonia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Congenital rubella infection (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Craniosynostosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exomphalos (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroschisis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genitalia external ambiguous (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Holoprosencephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypospadias (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Laryngomalacia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macrocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningomyelocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Micrognathia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multiple congenital abnormalities (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Multiple gastrointestinal atresias (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Persistent foetal circulation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 3 | 3 | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Necrotising colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6 | 3 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 4 | 4 | 3 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0 | 3 | 4 | 0 | 0
Sudden infant death syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | 3 | 2 | 0
Bartholin's abscess (Infections and infestations) | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 1
Bullous impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysentery (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 10 | 1 | 0 | 29 | 26 | 8 | 2
Giardiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 0 | 6 | 1 | 1 | 0
Malaria (Infections and infestations) | 9 | 6 | 4 | 0 | 4 | 9 | 3 | 1
Measles (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neonatal pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Neurosyphilis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmia neonatorum (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 5 | 2 | 1 | 0 | 7 | 5 | 0 | 0
Plasmodium malariae infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 5 | 0 | 0 | 34 | 33 | 8 | 6
Pneumonia bacterial (Infections and infestations) | 3 | 4 | 0 | 0 | 23 | 15 | 5 | 0
Post procedural sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Postpartum sepsis (Infections and infestations) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 3 | 0 | 0 | 1 | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Salmonella sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salpingitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 9 | 3 | 2 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 47 | 33 | 11 | 3
Sexually transmitted disease (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal scalded skin syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 12 | 8 | 4 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Wound sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Herbal toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine rupture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 5 | 0 | 0 | 1 | 1 | 0 | 0
Amniotic fluid volume decreased (Investigations) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foetal non-stress test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 22 | 20 | 11 | 2
Marasmus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Convulsion neonatal (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy neonatal (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 7 | 5 | 1 | 0 | 0 | 0 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 25 | 37 | 7 | 1 | 0 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 18 | 9 | 6 | 0 | 0 | 0 | 0 | 0
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 9 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 6 | 2 | 1 | 0
Labour pain (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 3 | 6 | 5 | 0
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 3 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 11 | 11 | 2 | 0 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 15 | 16 | 3 | 0 | 0 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 25 | 42 | 19 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 9 | 4 | 3 | 0 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 16 | 15 | 8 | 0 | 0 | 0 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 10 | 14 | 2 | 0 | 0 | 0 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 6 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 7 | 4 | 3 | 0 | 0 | 0 | 0 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 6 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 5 | 9 | 1 | 1 | 0 | 0 | 0 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brief psychotic disorder, with postpartum onset (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervix disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine atony (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Vulval haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 7 | 3 | 2 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 11 | 4 | 10 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 8 | 7 | 6 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 7 | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 5 | 4 | 2 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acrochordon excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection prophylaxis (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psychosocial support (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subgaleal haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mother, (AP) ZDV+sdNVP+TRV Tail (N=1547) | Mother, (AP) Triple ARV (3TC-ZDV/LPV-RTV) (N=1545) | Mother, (AP) Triple ARV (FTC-TDF/LPV-RTV) (N=445) | Mother, LP (N=204) | Infant, (Mother Received ZDV+sdNVP+TRV Tail) (N=1500) | Infant, (Mother Received Triple ARV (3TC-ZDV/LPV-RTV)) (N=1478) | Infant, (Mother Received Triple ARV (FTC-TDF/LPV-RTV)) (N=429) | Infant, LP (N=204)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 34 | 33 | 3 | 10 | 96 | 81 | 6 | 18
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 93 | 89 | 34 | 4
Eye discharge (Eye disorders) | 7 | 6 | 2 | 0 | 99 | 94 | 11 | 13
Abdominal pain (Gastrointestinal disorders) | 167 | 164 | 21 | 9 | 12 | 14 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 179 | 202 | 41 | 5 | 307 | 317 | 52 | 16
Gastritis (Gastrointestinal disorders) | 72 | 63 | 24 | 13 | 2 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 81 | 90 | 19 | 4 | 107 | 106 | 19 | 6
Pyrexia (General disorders) | 118 | 92 | 26 | 4 | 260 | 240 | 48 | 18
Body tinea (Infections and infestations) | 81 | 84 | 18 | 9 | 80 | 74 | 12 | 8
Conjunctivitis (Infections and infestations) | 37 | 30 | 10 | 6 | 99 | 75 | 20 | 8
Gastroenteritis (Infections and infestations) | 111 | 101 | 25 | 21 | 227 | 205 | 58 | 38
Malaria (Infections and infestations) | 85 | 79 | 17 | 4 | 103 | 95 | 29 | 2
Ophthalmia neonatorum (Infections and infestations) | 0 | 0 | 0 | 0 | 61 | 71 | 11 | 15
Oral candidiasis (Infections and infestations) | 13 | 8 | 0 | 1 | 124 | 112 | 44 | 14
Otitis media acute (Infections and infestations) | 10 | 11 | 8 | 1 | 74 | 62 | 30 | 2
Pharyngitis (Infections and infestations) | 88 | 92 | 21 | 12 | 37 | 35 | 5 | 4
Plasmodium falciparum infection (Infections and infestations) | 70 | 75 | 14 | 3 | 103 | 95 | 11 | 4
Pneumonia bacterial (Infections and infestations) | 18 | 25 | 2 | 6 | 94 | 84 | 25 | 5
Urinary tract infection (Infections and infestations) | 177 | 154 | 52 | 2 | 8 | 15 | 8 | 0
Vulvovaginal candidiasis (Infections and infestations) | 229 | 206 | 68 | 14 | 2 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 470 | 493 | 116 | 36 | 106 | 66 | 12 | 14
Aspartate aminotransferase increased (Investigations) | 68 | 88 | 29 | 12 | 4 | 3 | 0 | 1
Blood albumin decreased (Investigations) | 61 | 85 | 50 | 8 | 5 | 5 | 3 | 0
Haemoglobin decreased (Investigations) | 764 | 791 | 191 | 103 | 1226 | 1230 | 356 | 124
Hormone level abnormal (Investigations) | 25 | 30 | 11 | 15 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 668 | 619 | 161 | 67 | 859 | 848 | 255 | 115
Platelet count decreased (Investigations) | 151 | 144 | 41 | 18 | 94 | 94 | 40 | 9
Weight decreased (Investigations) | 112 | 85 | 21 | 10 | 29 | 20 | 16 | 2
White blood cell count decreased (Investigations) | 66 | 54 | 15 | 12 | 12 | 4 | 3 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 53 | 40 | 14 | 14
Growth failure (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 63 | 72 | 38 | 4
Headache (Nervous system disorders) | 189 | 188 | 23 | 8 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 272 | 271 | 52 | 26 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 80 | 78 | 9 | 1 | 2 | 1 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 116 | 136 | 21 | 5 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 179 | 173 | 20 | 6 | 274 | 253 | 35 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 13 | 2 | 0 | 78 | 80 | 30 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 81 | 93 | 12 | 1 | 144 | 138 | 23 | 8
Rash (Skin and subcutaneous tissue disorders) | 64 | 69 | 8 | 1 | 139 | 130 | 20 | 5
Rash generalised (Skin and subcutaneous tissue disorders) | 35 | 31 | 2 | 1 | 73 | 74 | 15 | 2
Hypertension (Vascular disorders) | 119 | 120 | 27 | 18 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights